CLINICAL TRIAL: NCT03003091
Title: Needs-Based Patient Education Versus Traditional Patient Education in Reducing Pre-operative Anxiety in Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulabhorn Hospital (Other)
Responsible Party: Principal Investigator, Apinut Wongkietkachorn, Doctor, Chulabhorn Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Chulabhorn
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Educational Problems; Surgery

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Needs-based patient education (Experimental): The participants received self-administered questionnaire to choose what topics they wanted to know and how much information they would like to know. After completing the questionnaire, the participants submit the questionnaire to their physicians (investigators). The surgeon then provided patient education based on participant needs.
  Interventions: Other: Needs-based patient education
- Traditional patient education (Active Comparator): The participants received all structured information
  Interventions: Other: Traditional patient education

INTERVENTIONS:
Other: Needs-based patient education
  Arms: Needs-based patient education
Other: Traditional patient education
  Arms: Traditional patient education

SUMMARY:
In patient education, the amount of information that is not proper with the individual patient, such as too much or too little, can increase anxiety to patient. Needs-based patient education has been developed to determine the proper amount of information and provide the education based on patient needs. This study aims to compare needs-based patient education to traditional patient education in how they affect preoperative anxiety and patient satisfaction.

DETAILED DESCRIPTION:
Preoperative anxiety can compromise surgical outcome. Anxiety increases serum cortisol, adrenaline, and noradrenaline. This results in postoperative pain, increased postoperative analgesic requirements, prolonged hospital stay and patient dissatisfaction. However, this anxiety can be reduced.

Patient education has been widely used to reduce operative anxiety; however, some patients have more anxiety after patient education. This incident could be explained by different individual's coping styles that patients use to deal with their anxiety. There are four major coping style: vigilant, avoidant, fluctuating, and flexible. Vigilant coper desires extended information to reduce anxiety. Avoidant coper desires minimal amount of information as too much will cause anxiety. Fluctuating coper generally desires small amount of information but desires greater detail in certain area. Flexible coper is able to adapt to whatever information available. Thus, if patient education with extended information is given to patients with avoidant coping style, they will have more anxiety. One study found that avoidant coping style is 31% of surgical patients in the study population. This is also supported by another study that one-third of patients reported to be worried after receiving an informative booklet. Therefore, to be able to deal with all types of coping style, patient education with different levels of information regarding patient needs is proposed to be developed.

Needs-based patient education has become more promising with increased supporting literature. It uses the principle of shared decision making, which is the pinnacle of patient-centered care. Needs-based patient education is also consistent with adult learning theory, which learning should be matched with different individual background and needs. A randomized controlled trial was conducted to compare needs-based patient education with traditional patient education in rheumatoid arthritis and found a superior result. However, there is still lack of evidence in using needs-based patient education in surgery.

This study evaluates needs-based patient education in reducing preoperative anxiety. To assess patient needs, a questionnaire is used as a tool. After receiving completed questionnaire, the physician provides information based on patient needs. Not only patients will benefit from this questionnaire but also physicians. The questionnaire enables physician to cut unnecessary information and pay more attention to the fact that patients need. Less information needed is less time spent in patient education session. As the most important reason why patient education is omitted is shortness of time. This needs-based patient education can contribute tremendously to the way we educate surgical patients.

Objectives This study aims to compare needs-based patient education to traditional patient education in how they affect preoperative anxiety, patient satisfaction, and time consumption.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* scheduled for day surgery
* willing to cooperate with the study

Exclusion Criteria:

* illegibility which could not answer questionnaire by themselves
* psychiatric diseases
* undergoing previous surgery within 6 months
* possibility to undergo major operation after day surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient anxiety before patient education (STAI) | 1 day
  Patient anxiety was assessed with Spielberger state-trait anxiety inventory (STAI)
Patient anxiety before patient education (VAS) | 1 day
  Patient anxiety was assessed with a 100 mm visual analogue scale for anxiety (VAS-anxiety)
Patient anxiety after patient education (STAI) | 1 day
  Patient anxiety was assessed with Spielberger state-trait anxiety inventory (STAI)
Patient anxiety after patient education (VAS) | 1 day
  Patient anxiety was assessed with a 100 mm visual analogue scale for anxiety (VAS-anxiety)
Patient anxiety after operation (STAI) | 1 day
  Patient anxiety was assessed with Spielberger state-trait anxiety inventory (STAI)
Patient anxiety after operation (VAS) | 1 day
  Patient anxiety was assessed with a 100 mm visual analogue scale for anxiety (VAS-anxiety)

SECONDARY OUTCOMES:
Patient Satisfaction before patient education | 1 day
  Patient satisfaction was measured by a 100 mm visual analogue scale.
Patient Satisfaction after patient education | 1 day
  Patient satisfaction was measured by a 100 mm visual analogue scale.
Patient Satisfaction after surgery | 1 day
  Patient satisfaction was measured by a 100 mm visual analogue scale.
Education time | 1 day
  Time in patient education was recorded with stopwatch at the beginning to the end of patient education session

REFERENCES:
- [Derived] Wongkietkachorn A, Wongkietkachorn N, Rhunsiri P. Preoperative Needs-Based Education to Reduce Anxiety, Increase Satisfaction, and Decrease Time Spent in Day Surgery: A Randomized Controlled Trial. World J Surg. 2018 Mar;42(3):666-674. doi: 10.1007/s00268-017-4207-0. PMID 28875242